CLINICAL TRIAL: NCT04673825
Title: Effectiveness and Cost-effectiveness of Monitoring Spondyloarthritis With the Integrated eHealth System SpA-Net: a Randomized Controlled Trial
Brief Title: Monitoring Spondyloarthritis With SpA-Net
Acronym: TeleSpA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other); Medisch Spectrum Twente (Other); Dutch Arthritis Association (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NL71041.068.19
Record Dates: First submitted 2020-12-01; First posted 2020-12-17 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Spondyloarthritis; Ankylosing Spondylitis; Psoriatic Arthritis; Spondyloarthropathy
Keywords: Telemonitoring; Patient initiated care; Remote care; eHealth; Cost-effectiveness
MeSH Terms: conditions — Spondylarthritis; Spondylitis, Ankylosing; Arthritis, Psoriatic; Spondylarthropathies

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: patient initiated care + telemonitoring (Experimental): Patients in the intervention group will only have a scheduled outpatient visit at baseline and after 1 year. Patients will answer questionnaires and have routine blood tests done before every visit. At 6 months, there will be a remote monitoring check-up and results will be checked by the physician. If indicated, a telephone or video call can take place or a physical visit can be planned. Patients from either arm will be instructed that at any time, they may contact the rheumatology department and extra visits can be scheduled. During the COVID-pandemic, outpatient visits may also take place through telephone or video calls.
  Interventions: Other: Patient initiated care + telemonitoring
- Control group (No Intervention): The standard care group will have a scheduled outpatient visit at baseline and after 1 year, and in between as usual, scheduled at the discretion of the treating rheumatologist. Prior to each visit, patients complete questionnaires in SpA-Net and have routine blood tests done. Patients from either arm will be instructed that at any time, they may contact the rheumatology department and extra visits can be scheduled. During the COVID-pandemic, outpatient visits may also take place through telephone or video calls.

INTERVENTIONS:
Other: Patient initiated care + telemonitoring — See arm/group descriptions.
  Arms: Intervention: patient initiated care + telemonitoring

SUMMARY:
Randomized controlled trial to assess the effectiveness and cost-effectiveness of an intervention combining patient initiated care and telemonitoring through the online eHealth platform SpA-Net versus standard care for patients with spondyloarthritis.

DETAILED DESCRIPTION:
Multicenter randomized controlled trial to investigate the effectiveness and cost-effectiveness of telemonitoring through SpA-Net, in combination with patient initiated care, versus standard care. Participants will be recruited at the outpatient clinics of participating centers, and will be randomised (after informed consent) into either the telemonitoring or standard care group. Patients in both arms will use SpA-Net and will be followed up for 1 year. Concomitantly a trial-based cost-utility analysis will be performed.

Randomisation (1:1; intervention versus standard care) is done using the minimisation method, stratifying for medical centre, subtype of SpA (axial, peripheral or combined) and treatment (biological use versus no biological use). Due to the nature of the intervention neither patients nor clinicians can be blinded to the allocation.

A sample size of 80 patients per group is necessary to detect the primary outcome with a power of 0.80 and alpha of 0.05. Assuming a 20% drop-out during follow-up, 100 patients per group will be included. This sample size also suffices to show non-inferiority for all secondary objectives with a power of 0.80 and a one-sided alpha of 0.025.

Study endpoints

A. The primary endpoint is defined as at least 25% reduction in the number of rheumatology department outpatient visits in the intervention group compared to the standard care group, within a 1-year follow-up period. Due to the COVID-19 pandemic these may also take place through telephone or video calls, replacing physical visits.

B. Secondary study parameters/endpoints

* Non-inferiority of telemonitoring compared to standard care with respect to quality of care and health outcomes.
* Non-inferiority with respect to experience with SpA-Net and general rheumatological care.
* Association between patient-reported self-management skills and successful application of telemonitoring
* Experience with telemonitoring through SpA-Net among care providers
* Difference between the populations with regard to healthcare cost per quality adjusted life year (QALY) gained after 1 year
* Difference between the populations with regard to societal cost per QALY gained after 1 year

STATISTICAL ANALYSIS The primary outcome will be analysed in the intention to treat (ITT) population. The differences between the two groups with respect to quality of care aspects and overall resource utilisation will be analysed in the ITT and the per-protocol (PP) population. All other secondary outcomes will be analysed in the ITT population.

The primary endpoint will be compared between both groups with ANOVA. Given that the population is randomised, an equal distribution of baseline characteristics is to be expected. In case differences between the two groups exist on baseline (visually), post-hoc analyses adjusting for these differences will be done (ANCOVA).

Secondary endpoints will be analysed with ANOVA. Post-hoc, subgroup analyses and predictive analyses with respect to self-management skills and and successful application of telemonitoring will be done with linear mixed-effect models with each endpoint as dependent variable and time, group and their interaction as fixed effects. Descriptive statistics will be used to summarize experience with telemonitoring among care providers.

Non-inferiority margins for secondary outcome measures:

* For ASDAS, non-inferiority is defined as an increase of no more than 0.9.
* A change in BASDAI of < 2.0 will be considered non-inferior.
* A cut-off of 20 millimetres is used for the patient global VAS, and a cut-off of 10 millimetres for the physician global VAS.
* An increase in VAS pain of no more than 20 millimetres will be considered non-inferior.
* At the time of the study proposal, approximately 90% of the patients is satisfied with the care provided. Non-inferiority is defined as a decrease of no more than 5%.

Health economic evaluation will be performed in accordance with the ISPOR guidelines, as well as the current Dutch guidelines for economic evaluations in healthcare. Analyses will be done both from a Dutch healthcare and societal perspective.

Currently, no consensus exists with regard to disease weights for SpA. As such, results will be reported for willingness-to-pay thresholds of both 20.000 and 50.000 euros per QALY gained. Sensitivity analyses will be performed to test the robustness of the results gathered.

Missing data will be addressed using multiple imputation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18+ years)
* Diagnosis of SpA according to treating physician
* At least 2 years of disease duration, to be familiar with signs, symptoms, and medication
* Stable disease, defined as being in a patient acceptable symptom state according to patient AND treating physician AND no treatment change expected in the next few months
* Access to a computer, tablet and/or smartphone for the entire duration of the study

Exclusion Criteria:

* Insufficient mastery of Dutch language
* Incompetent to act for oneself
* Limited life expectancy
* Ongoing (or planned) pregnancy during the study period
* Patients participating in other research project(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Number of scheduled and unscheduled outpatient visits to the rheumatology department. | 1 year
  Comparison of total number of outpatient visits in a 1-year period between intervention and control group.

SECONDARY OUTCOMES:
Ankylosing Spondylitis Disease Activity Score (ASDAS) | 1 year
  ASDAS is a composite index to assess disease activity in ankylosing spondylitis. Parameters included are C-reactive protein value (mg/L) and four self-reported items (0-10, numerical rating scale [NRS]): back pain, duration of morning stiffness, peripheral pain/swelling and patient global assessment of disease activity. Higher scores on individual parameters represent more severe symptoms. Higher ASDAS represents higher disease activity.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 1 year
  BASDAI consists of 6 questions representing the 5 major symptoms of ankylosing spondylitis (AS), every question is answered by using a 0-10 numerical rating scale with higher scores representing more severe symptoms: fatigue, spinal pain, joint pain / swelling, areas of localized tenderness, morning stiffness duration, morning stiffness severity. The mean of the two scores relating to morning stiffness is taken. The resulting sum of all scores (0 to 50 score) is divided by 5, resulting in a 0 - 10 BASDAI score, with increasing scores representing more active disease.
Global well-being patient | 1 year
  Assesses the patient's global well-being during the last week on a Visual Analogue Scale, range: 0-100 mm. A score of 100 mm represents the worst outcome.
Patient reported pain | 1 year
  Visual Analogue Scale, 0-100 mm. A score of 0 equals no pain. Higher scores represent more severe pain.
Disease activity according to physician | 1 year
  Visual Analogue Scale, 0-100 mm. A score of zero equals no disease activity. Higher scores represent more active disease.
C-Reactive Protein (CRP) | 1 year
  Amount of CRP detected in blood samples, expressed in mg/L.
Tender Joint Count 66 / Swollen Joint Count 68 | 1 year
  Only if present, the number of tender (0-66) and swollen (0-68) joints will be evaluated by an independent assessor at each physical outpatient visit.
Presence of dactylitis and/or enthesitis | 1 year
  If present, dactylitis (presence/absence, locations) and enthesitis (presence/absence, locations) will be evaluated by an independent assessor at each physical outpatient visit.
Psoriasis severity: Body Surface Area (BSA) | 1 year
  Measurement of total area of patient's body affected by psoriasis, expressed in percentages (range: 0 - 100).
Psoriasis severity: Nail involvement | 1 year
  Nail changes due to psoriasis will be reported as either present (yes) or absent (no).
36-item Short Form Health Survey (SF-36) | 1 year
  The SF-36 survey contains 36 items, covering eight domains and one single item that provides an indication of perceived change in health. Aggregate percentage scores will be calculated for two components (Mental Component Score [MCS] and Physical Component Score [PCS]). Range: 0% (worst possible level of functioning) to 100% (best possible level of functioning).
EuroQol with 5 dimensions and 5 point Likert scale (EQ-5D-5L) | 1 year
  The EQ-5D-5L evaluates five dimensions, each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, extreme problems). This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. In addition, a vertical Visual Analogue Scale records the patient's self-rated health (range: 'The worst health you can imagine' [0 mm, bottom-end] to 'The best health you can imagine' [100 mm, top-end]).
Assessment of SpondyloArthritis international Society health index (ASAS HI) | 1 year
  The ASAS HI contains 17 dichotomous response items (0 = 'I do not agree'; 1 = 'I agree'). A sum score is calculated, resulting in a total ASAS HI score ranging from 0 to 17. Lower scores indicate a better health status.

OTHER OUTCOMES:
Healthcare cost per quality adjusted life year (QALY) gained after 1 year | 1 year
  Self-reported health resource utilisation will be evaluated for two separate 6-month recall periods. Total resource consumption will be reported as the sum of resources utilized during the entire 12-month study period.
Societal cost per QALY gained after 1 year | 1 year
  To calculate societal costs, self-reported professional absenteeism will be used. Paid productivity loss is valued using the friction cost method as per Dutch national guidelines with a friction period of 85 days. Presenteeism (decreased productivity while at work due to illness) and unpaid productivity loss will be measured and valued based on Dutch costing guidelines.
Quality Adjusted Life Years (QALY) | 1 year
  To determine incremental cost-utility (iCU), utility will be measured in QALYs. Results from health-related quality of life measures will be converted into utility scores (0-1) to allow calculation of QALYs. Where available, Dutch tariffs will be used.
Self-management characteristics | Baseline
  As measured by the Self-Management Screening questionnaire (SeMaS) which contains 27 items, assessing a total of 10 domains. Each domain has three possible scores (low = important barrier for self management, middle = unclear/possible barrier for self management, high = self-management likely to be successful). Different combinations of scores result in different patient profiles.
Experience with telemonitoring through SpA-Net among care providers | 1 year
  Global satisfaction and agreement on statements (safety, effectiveness, patient-centeredness, timeliness, efficiency, equitability, flexibility, use of time and resources) about telemonitoring with SpA-Net, measured on a 5 point Likert scale (range: 'I strongly agree' to 'I strongly disagree').

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Medisch Spectrum Twente, Enschede, Overijssel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hermans K, Webers C, Boonen A, Vonkeman HE, van Tubergen A. Patient-initiated follow-up supported by asynchronous telemedicine versus usual care in spondyloarthritis (TeleSpA-study): a randomised controlled trial of clinical and cost-effectiveness. Lancet Rheumatol. 2024 Dec;6(12):e848-e859. doi: 10.1016/S2665-9913(24)00229-7. Epub 2024 Nov 1. PMID 39492125
- [Derived] Hermans K, Boonen A, Vonkeman HE, van Tubergen A. Effectiveness and cost-effectiveness of combined asynchronous telemonitoring and patient-initiated care for spondyloarthritis: protocol for a pragmatic multicentre randomised controlled trial (TeleSpA Study). BMJ Open. 2023 Feb 20;13(2):e067445. doi: 10.1136/bmjopen-2022-067445. PMID 36806136